CLINICAL TRIAL: NCT03691051
Title: Pyrotinib Plus Capecitabine in Patients With Brain Metastases From HER2-positive Metastatic Breast Cancer : a Single-arm, Open-label, Ahead Study
Brief Title: A Study of Pyrotinib Plus Capecitabine in Patients With Brain Metastases From HER2-positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-MBC-HN001
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: HER2 Positive Metastatic Breast Cancer
MeSH Terms: interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib Plus Capecitabine (Experimental): Pyrotinib + Capecitabine
  Interventions: Drug: Pyrotinib plus Capecitabine

INTERVENTIONS:
Drug: Pyrotinib plus Capecitabine — Pyrotinib:400mg/d,q.d.,p.o. A course of treatment need 21days. Capecitabine:1000mg/m2,bid,from day1-day14, A course of treatment need 21 days.
  Other Names: Irene

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors.This study is a single-arm, prospective, open label clinical study of pyrotinib plus capecitabine as the Therapy of brain metastases from HER2-positive metastatic breast cancer.

DETAILED DESCRIPTION:
Brain metastases occur in 30-50% of patients with metastatic HER2-positive breast cancer. In the case of solitary brain metastases, surgery or stereotactic radiosurgery are the preferred therapeutic approaches.Chemotherapy is used after further progression of disease but it has limited effectiveness. In HER2-positive tumours, trastuzumab therapy has been postulated to be associated with an increased risk of development of brain metastases.Thus new therapeutic options are urgently needed to improve patients'outcome. Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER-1 and HER-2 receptors. We designed the study to explore the possibility of pyrotinib plus capecitabine for brain metastases from HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years old at the time of signing the informed consent form.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
3. HER2-positive: In the pathological examination/rechecking of primary lesions or metastatic lesions performed by the Research site's Pathology Laboratory, at least once the tumor cells defined as 3+ staining by immunohistochemistry, or fluorescence in situ hybridization [FISH] confirmed positive
4. MRI/enhanced CT confirmed brain metastasis. According to RECIST 1.1, there is at least one measurable brain lesion, and the measurability of extracranial lesions is not required
5. Patients Group Cohort A: participants with brain metastases who have not previously been treated with CNS radiotherapy, it should be more than two weeks since the end of the last systemic treatment. Patients with new brain lesions after craniotomy are allowed to be included, provided that they have not received radiotherapy after surgery and are at least 2 weeks away from surgery.

   Cohort B: Patients with disease progression or new lesions after whole brain radiotherapy (WBRT) or stereotactic radiotherapy (SRT); For lesions that have received local treatment, there is clear evidence of progress in imaging examination, and the lesions that have undergone radiotherapy can be selected as target lesions. If a patient has multiple CNS lesions, only one or a few of which are treated with SRT, and there are lesions that are not treated locally, such patients are still eligible for enrollment in this study.
6. Previous treatment

   Acceptable previous treatments:

   History of trastuzumab and other anti-HER2 macromolecular antibodies. Any lines of previous chemotherapy. History of endocrine therapy. Patients who have not used capecitabine except for patients with progression at least 6 (for metastatic disease) or 12 (as adjuvant therapy) months after discontinuation of a capecitabine-containing treatment.

   Concurrent use of bisphosphonates, mannitol and glucocorticoids is allowed, provided that the dosage(⩽2 mg dexamethasone (or equivalent) per day) of glucocorticoids is stable for at least one week before enrollment.
7. Expected to survival ≥ 6 months
8. Patients must have adequate organ function, criteria as follows.

   1. Blood routine examination：Absolute Neutrophil Count (ANC)≥1.0×109/L； PLT ≥100×109/L； Hb ≥90g/L
   2. Blood chemistry test：TBIL ≤1.5 times the upper limit of normal (ULN); ALT and AST≤3 times ULN; For patients with liver metastases, ALT and AST≤5×ULN; BUN and Cr≤1×ULN and creatinine clearance ≥50mL/min (CockcroftGault formula);
   3. Ultrasonic cardiogram: LVEF≥50%
   4. 12-lead ECG: The QT interval (QTcF) corrected by Fridericia's method is < 450 ms/man and < 470 ms/women.
9. Patients need to voluntarily join this study after they fully understand and sign the informed consent form. Patients need to have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients with leptomeningeal metastasis (diagnosed by imaging/positive cerebrospinal fluid cytology) or a clear indication of clinically significant leptomeningeal involvement;
2. CNS complications that require urgent neurosurgical intervention (e.g. resection, shunt placement). Patients with poorly response brain metastases after dehydration treatment and glucocorticoid treatment. Such as uncontrollable increase in intracranial pressure, jet vomiting, mental disorders, epilepsy, cognitive impairment, etc.
3. Third space fluid that cannot be controlled by drainage or other methods (such as large amounts of pleural fluid and ascites);
4. Patients who have received chemotherapy, surgery or molecular targeted therapy within 2 weeks before enrollment; patients who have received endocrine therapy within 1 week before enrollment; minor surgery, such as tumor biopsy, thoracentesis or intravenous catheterization or the like are allowed;
5. Participated in other clinical trial within 4 weeks prior to randomization.
6. Concurrent treated, or who has been treated with HER2 tyrosine kinase inhibitors (including lapatinib, neratinib, pyrotinib, etc.);
7. History of other malignant tumors within 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma;
8. Receiving any other anti-tumor therapies at time of study screening visit.
9. There are serious and/or uncontrolled complications that may affect participation, including any of the following:

   1. dysphagia, chronic diarrhea and intestinal obstruction and factors that affect the administration and absorption of the drug;
   2. Allergic constitution; Allergic to the study drug; History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency diseases; History of organ transplantation;
   3. History of severe heart disease, including: myocardial infarction and heart failure; any other heart disease that is not suitable for participation (investigator assessment);
   4. Infection.
10. Female patients during pregnancy and lactation; fertile female patients who tested positive on a baseline pregnancy test; female patients of childbearing age who are unwilling to take effective contraceptive measures during the trial.
11. Any other circumstances that are not suitable for inclusion in this study (investigator assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate of Intracranial Lesion (ORR) | Estimated up to 1 year
  the proportion of patients with the best intracranial response of confirmed complete or partial response according to RECIST 1·1, as assessed by the investigator

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Estimated up to 3 year
  time from the first dose to disease progression or any-cause death
Objective Response Rate of Extracranial Lesion (ORR) | Estimated up to 1 year
  proportion of patients with confirmed extracranial complete or partial response per RECIST 1·1
Duration of response (DOR) | Estimated up to 1 year
  time from the first documented intracranial objective response to intracranial or extracranial disease progression in patients with confirmed response
Overall survival（OS） | Estimated up to 3 year
  time from the first dose of study drug to any-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identificationare available following article publication.
Supporting Information: Study Protocol
Time Frame: Three years from publication
Access Criteria: Please contact Central contact person by Email

REFERENCES:
- [Derived] Yan M, Ouyang Q, Sun T, Niu L, Yang J, Li L, Song Y, Hao C, Chen Z, Liu Z, Lv H, Zhang M, Liu L, Yang X, Xiao H, Gao Z, Li X, Dong F, Zhang L, Dong D, Chen X, Qiao J, Zhang G, Zeng H, Wang J, Sun H, Feng Y, Chen Y, Xia F. Pyrotinib plus capecitabine for patients with HER2-positive metastatic breast cancer and brain metastases (PERMEATE trial): overall survival results from a multicenter, single-arm, two-cohort, phase 2 trial. EClinicalMedicine. 2024 Sep 20;76:102837. doi: 10.1016/j.eclinm.2024.102837. eCollection 2024 Oct. PMID 39380967
- [Derived] Yan M, Ouyang Q, Sun T, Niu L, Yang J, Li L, Song Y, Hao C, Chen Z, Orlandi A, Ishii N, Takabe K, Franceschini G, Ricci F, Verschraegen C, Liu Z, Zhang M, Lv H, Liu L, Yang X, Xiao H, Gao Z, Li X, Dong F, Chen X, Qiao J, Zhang G. Pyrotinib plus capecitabine for patients with human epidermal growth factor receptor 2-positive breast cancer and brain metastases (PERMEATE): a multicentre, single-arm, two-cohort, phase 2 trial. Lancet Oncol. 2022 Mar;23(3):353-361. doi: 10.1016/S1470-2045(21)00716-6. Epub 2022 Jan 31. PMID 35085506